CLINICAL TRIAL: NCT06745258
Title: ICARE-LCS QUERI Partnered Evaluation Initiative: Integrating Comprehensive Tobacco Treatment to Enhance Lung Cancer Screening (PEC 24-239)
Brief Title: ICARE-LCS QUERI Partnered Evaluation Initiative: Integrating Comprehensive Tobacco Treatment to Enhance Lung Cancer Screening
Acronym: ICARE-LCS
Status: Not yet recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Oncology and Precision Medicine (Unknown); VA Tobacco Use Treatment National Program Office (Unknown); VA National Center for Lung Cancer Screening (Unknown)
Responsible Party: Sponsor
Other Study IDs: PEX 24-002
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Dependence Treatment; Lung Cancer Screening
Keywords: Lung Cancer; Lung Nodule; Tobacco; Lung Cancer Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Veterans Participating in Lung Cancer Screening who Smoke: Veterans participating in lung cancer screening who smoke and are receiving care at participating VA medical centers
- Participating VA Medical Centers: Seven sites that have agreed to participate in implementation intervention
  Interventions: Other: External Facilitation

INTERVENTIONS:
Other: External Facilitation — Multi-component facilitation strategy to address identified implementation needs
  Groups: Participating VA Medical Centers

SUMMARY:
Lung cancer is the leading cause of cancer-related death among Veterans with 90% of cases attributable to smoking. Lung cancer screening (LCS) combined with smoking cessation saves the most lives. ICARE-LCS seeks to decrease health inequality and improve Veteran health by reducing smoking rates among Veterans receiving LCS. ICARE-LCS will use implementation methods to inform national cancer prevention efforts and build infrastructure necessary to support broad implementation of high-impact tobacco dependence treatment (TDT) processes in LCS programs.

DETAILED DESCRIPTION:
The primary goal is to improve the delivery of tobacco dependence treatment (TDT) within Veterans Affairs (VA) lung cancer screening (LCS) programs. LCS with annual low-dose computed tomography saves lives through the early detection of lung cancer and is being broadly deployed, now at 113 VA medical centers. Due to the eligibility criteria selecting for current or previous smoking, 50-60% of LCS participants currently smoke. Modeling studies support that integrating TDT into LCS nearly doubles the benefit of the screening itself. Therefore, access to high-quality TDT is a program requirement per the VA LCS guidance memo.

Though a robust integration of LCS and TDT is a VA priority, in reality there remains a gap in both reach and intensity of TDT for LCS participants. Guidelines and evidence support TDT processes that include 1) systematic assessment and connection to treatment (e.g. Ask-Advise-Connect, motivational interviewing, optout or proactive strategies) and 2) treatment that includes the evidence-based combination of intensive pharmacologic and behavioral treatments ('combined TDT'). Recent trials in LCS participants found high rates of agreeing to treatment using 'opt-out' motivational referral strategies and the highest cessation rates using a longitudinal "chronic disease" model that delivers combined TDT over a period up to a year. Unfortunately, relatively few Veterans in LCS receive any TDT and the treatment is usually inconsistent with guidelines and this evidence. In a national sample of LCS participants who smoke, only 16.4% received any pharmacotherapy for TDT, many under-dosed with short-acting nicotine replacement alone, and fewer than 1% received the recommended combination of behavioral and pharmacologic treatment. This represents a significant gap in care. Improving quality of TDT for Veterans in LCS has been identified as a priority area by multiple stakeholders including the Office of Oncology and Precision Medicine (OPM), the investigators' operational partner, the VA Lung Precision Oncology Program (LPOP), the White House Prevention and Screening Task Force, the National Committee for Quality Assurance and Veterans engagement groups. Each care process-LCS and TDT-is complex on its own, which has hampered integration. While some LCS processes are standardized across VA through use of the tools provided by the National Center for Lung Cancer Screening (NCLCS), individual LCS programs use varied care models. Programs can be 'centralized' (most LCS-related care is delivered by dedicated program staff) or 'hybrid,' where responsibilities are shared between primary care and LCS staff. NCLCS has worked with VAs across the country to enhance LCS quality and uptake. Individual LCS programs deliver combined TDT variably, and many processes are not adapted for the longitudinal, annual LCS process. The VA Tobacco Use Treatment Program Office (TUT) is currently conducting a pilot funded by the Cancer Moonshot to demonstrate feasibility of integrating TDT into LCS, recently expanded from 11 to 15 sites. The Minneapolis VA has conducted a VISN 23-Quality Enhancement Research Initiative (QUERI) partnered implementation pilot to understand barriers and needs among diverse LCS programs, identifying many modifiable targets. The VISN 23 QUERI Team and TUT have collaborated to design an LCS-TDT toolkit that will soon be nationally available. While an important step, a toolkit alone may be insufficient to increase uptake of best practices. Tailored implementation support through intensive external facilitation may be necessary to effectively integrate TDT processes within the VA LCS landscape. With support from the operational partner, OPM, this project proposes to work with TUT and the NCLCS to build on existing efforts to increase participation in combined TDT for LCS participants. This project will utilize both retrospective data analysis and prospective data gathering to inform and tailor a toolkit for national dissemination. ICARE-LCS is an implementation evaluation study model.

Specific Aims:

Aim 1: Identify key process components of effective tobacco treatment programs in LCS and success factors for providing combined TDT. A mixed methods assessment will be conducted at 10 sites in the TUT Moonshot pilot, first qualitatively assessing their current TDT-LCS processes, success factors and perceived barriers to implementation of combined TDT. Data will then be linked with quantitative data of treatment participation and short-term cessation. Findings will be used to refine the toolkit for use in Aim 2 and nationally.

Aim 2: Test a multicomponent facilitation package to improve integration of TDT and LCS.

Seven programs will be identified from among LPOP sites outside of the TUT pilot, ensuring variation in site characteristics (e.g. hybrid vs centralized model), and provided implementation support using external facilitation. Sites will be matched at least 1:1 to another site in the LPOP network that will receive implementation as usual (controls). The primary outcome will be penetration (participation in combined TDT, secondary outcome any treatment) with additional secondary outcomes of fidelity (ideal TDT), and effectiveness (short-term cessation).

Aim 3: Evaluate the implementation outcomes of feasibility, acceptability, fidelity, appropriateness, and cost of implementing TDT integrated with LCS, assessed among Veterans and care team members.

Implementation outcomes other than cost will be assessed using qualitative methods. Cost will be examined related to the implementation support and to the TDT provided (e.g. LCS staff costs, pharmacotherapy, tobacco-related visits) using staff logs and VA pharmacy and billing data. Collectively, the above program evaluation will inform national cancer prevention efforts and build infrastructure necessary to support broad implementation of high-impact TDT processes in LCS programs.

ELIGIBILITY:
Inclusion Criteria:

This is a VAMC based Quality Improvement Partnered Evaluation Initiative. VA sites from around the country that agreed to participate are included.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating VA Medical Centers
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Receipt of Combined Tobacco Dependence Treatment | Approximately 3 years
  Participation in counseling and pharmacotherapy within 90 days of lung cancer screening referral

SECONDARY OUTCOMES:
Number of Veterans Receiving ANY Tobacco Dependence Treatment Therapy | Approximately 3 years
  Participation in ANY tobacco dependence treatment therapy (including but not limited to pharmacotherapy or counseling) for eligible Veterans in lung cancer screening who smoke
Number of Veterans Receiving of Pharmacotherapy or Counseling Alone | Approximately 3 years
  Participation in individual treatment options among patients in lung cancer screening who smoke. These are defined as Pharmacotherapy (nicotine replacement, bupropion, varenicline, combination treatments) and counseling (individual or group tobacco visits delivered by any modality).
Cost Associated with Tobacco Dependence Treatment Among Lung Cancer Screening Participants who Smoke | Approximately 3 years
  Evaluate facility level costs and economic impacts of tobacco treatment for patients in lung cancer screening who smoke.
Rate of Short-term Cessation Among Veterans In Lung Cancer Screening who Smoke | Approximately 3 years
  Short-term cessation data among eligible Veterans in lung cancer screening who smoke as gathered by chart review
Implementation Outcomes Assessed at Participating Sites | Approximately 3 years
  Assessing implementation outcomes by qualitative review.

CONTACTS AND LOCATIONS:
Overall Officials: Anne C. Melzer, MD MS, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No